CLINICAL TRIAL: NCT02984800
Title: The Anesthetic and Analgesic Effectiveness of Single Paravertebral Blockade Injection for Herniorrhaphy in Children
Brief Title: Effectiveness of Single Paravertebral Blockade Injection for Herniorrhaphy in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Zoher Naja, Chairperson of Anesthesia and Pain Management Department, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 3122016
Record Dates: First submitted 2016-12-03; First posted 2016-12-07 (Estimated); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Reduce Pain After Herniorrhaphy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Group I (Experimental): Patients will receive one PVB injection at L1-L2 .
  Interventions: Other: Anesthesia induction; Other: PVB injection at L1-L2
- Group III (Experimental): Patients will receive three PVB injections at T12-L1, L1-L2 and L2-L3.
  Interventions: Other: Anesthesia induction; Other: PVB injections at T12-L1, L1-L2 and L2-L3.

INTERVENTIONS:
Other: Anesthesia induction — All patients will have inhaled induction of anesthesia by facemask using oxygen and 8% sevoflurane for 2 to 4 minutes followed by placement of an IV cannula. After performing PVB injections, the sevoflurane concentration will be decreased to 0.4% to 0.8% and maintained until completion of surgery.
Other: PVB injection at L1-L2 — Patients will receive a single PVB injection at L1-L2 and placebo PVB injections at T12-L1 and L2-L3.
  Arms: Group I
Other: PVB injections at T12-L1, L1-L2 and L2-L3. — Patients will have PVB injections at T12-L1, L1-L2 and L2-L3.
  Arms: Group III

SUMMARY:
Paravertebral block (PVB) might be a technique of choice for hernia surgery due to its unilateral segmental anesthesia of the operative site, good muscle relaxation and prolonged postoperative analgesia. Despite PVB effectiveness, a continuing search for a reliable, timely and effective technique generates the investigation of a single PVB injection for children undergoing unilateral inguinal hernia repair. Two theoretical concepts were behind this investigation. First, possible spread of single PVB injection in the lumbar area over dermatomes corresponding to the inguinal hernia region in children likewise the spread over multiple adjacent segments from a single thoracic PVB injection. Second, as the inguinal region receives innervation from the ilioinguinal, iliohypogastric and genitofemoral nerves, all three arising from L1-L2 level; thus, a single PVB injection at this level could provide unilateral segmental anesthesia.

DETAILED DESCRIPTION:
The study will be conducted prospectively, using a randomized double-blinded design. Male patients scheduled for elective unilateral herniorrhaphy will be included in the study.

Patients will be randomly allocated into two groups using the sealed envelope technique. All patients will have inhaled induction of anesthesia by facemask using oxygen and 8% sevoflurane for 2 to 4 minutes followed by placement of an IV cannula. After performing PVB injections, the sevoflurane concentration will be decreased to 0.4% to 0.8% and maintained until completion of surgery.

Then, group I will receive one PVB injection at L1-L2 and placebo PVB injections at T12-L1 and L2-L3. Group III will receive three PVB injections at T12-L1, L1-L2 and L2-L3.

Paravertebral block technique After induction of anesthesia and placement of regular anesthetic monitors, three unilateral PVBs will be performed with the child lying in the lateral position with the operative side uppermost. The needle insertion sites will be 1.5-2.0 cm lateral to the midline depending on the age and the body mass index of the child.

After aseptic preparation of the skin, a nerve stimulator (Stimuplex, B Braun AG, Melsungen, Germany) is used to identify an evoked muscular contraction appropriate for the levels. A 50 mm 21G insulated needle (Stimuplex A, B Braun AG) will be introduced perpendicular to the skin using 5 mA and 1 Hz. Then, the stimulating needle is gently manipulated to allow for adequate muscle response with a stimulating current of 0.4-0.6 mA.

In order to preserve the double-blindness of this trial, an independent nurse will prepare three syringes. Each syringe is labeled with the corresponding level of injection i.e, T12-L1, L1-L2 and L2-L3. The T12-L1 and L2-L3 syringes that will be used for group I will contain 0.45 ml placebo (0.9% normal saline) per syringe. The syringe labeled L1-L2 will contain 0.45 ml local anesthesia. On the other hand, the three syringes that will be used for group III will contain 0.15 ml local anesthesia and 0.3 ml placebo. Consequently, all patients will receive a total of 0.45 ml anesthesia and 0.9 ml placebo.

Data collection Demographic data such as age, weight and height will be collected. Non-invasive mean arterial blood pressure and heart rate will be recorded preoperatively (baseline), intraoperatively (incision of skin, dissection of hernia, traction over the sac and closure of incision) and immediately postoperatively. During the operation, any hemodynamic changes in excess of 15% from baseline values will result in a step-wise increase or decrease of the sevoflurane concentration. Intra-operative sevoflurane concentration will be recorded.

Postoperative pain assessment and analgesia As for pain assessment, the Face, Legs, Activity, Cry, Consolability (FLACC) scale will be used to measure postoperative pain (0 indicating no pain and 10 maximum possible pain).

Patients with pain score greater than 4 are given 1-2 mg/kg Tramadol hydrochloride (Tramal drops, Laboratoire Grunenthal, Aachen, Germany) A 350 mg paracetamol suppository (Tylenol CILAG SA, Schaffhouse, Switzerland) will be prescribed in pain score is less than 5.

During hospitalization trained nurses, blinded to the randomization, will collect the pain scores. Following hospital discharge, pain scores will be assessed by parents through phone calls made by the same nurses during the first postoperative day at predetermined time intervals (0h, 6h, 12h, 24h).

ELIGIBILITY:
Inclusion Criteria:

* elective unilateral herniorrhaphy

Exclusion Criteria:

* history of allergic reactions to local anesthetics
* bleeding diatheses
* spinal abnormality

Ages: 2 Months to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Analgesic consumption | 24 hours postoperatively
  Analgesics consumed will be recorded

SECONDARY OUTCOMES:
Hemodynamic stability | During the operation (approximately one hour)
  Hemodynamic stability measured through mean arterial pressure (MAP)

CONTACTS AND LOCATIONS:
Locations (1):
- Makassed General Hospital, Beirut, Lebanon